CLINICAL TRIAL: NCT05991492
Title: Improving Sleep With a Digital Cognitive Behavioral Therapy for Insomnia Application
Acronym: STELLAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Sogol Javaheri, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023P001950
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based Cognitive Behavioral Therapy for Insomnia (wCBT-I) with general sleep education (Active Comparator)
  Interventions: Device: Web-based Cognitive Behavioral Therapy for Insomnia (wCBT-I
- General Sleep Education (No Intervention)

INTERVENTIONS:
Device: Web-based Cognitive Behavioral Therapy for Insomnia (wCBT-I — Digital insomnia treatment
  Arms: Web-based Cognitive Behavioral Therapy for Insomnia (wCBT-I) with general sleep education

SUMMARY:
Insomnia is an important public health problem and the most common sleep disorder in the general population. Up to 20% of adults in the United States suffer from insomnia disorder, and it has been associated with increased morbidity, mortality, and healthcare costs. Cognitive behavioral therapy for insomnia (CBT-I) is the initial recommended treatment approach for insomnia. Combined therapy with CBT-I and medication has shown no advantage over CBT-I alone. CBT-I is not always accessible to patients, however, due to cost and availability of trained healthcare professionals. Web-based CBT-I is an inexpensive and effective self-management tool for treatment of insomnia.

This pilot study would test the efficacy of a new digital CBT-I application called Stellar Sleep, a cost effective and user-friendly version of wCBT-I, in patients with insomnia. This is the first digital CBT-I app that allows automatic entry of sleep diary data from wearable devices that track sleep (such as the Mi Band 5 or a FitBit, for instance). Testing the efficacy of this application will provide the preliminary data necessary for larger trials to further validate the application and determine its role for future patients. Use of this application can help bridge the gap in providing care to insomnia patients with transportation and cost barriers and to accommodate the long wait times for traditional in-person CBT-I. It will also be the first web-based CBT-I application that can directly upload data from a wearable device.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Daily access to a computer or smartphone with reliable internet connection

Exclusion Criteria:

* Currently pregnant or planning to become pregnant in the next year
* Visual impairment that prevents use of a computer
* Serious health conditions that will prevent taking part in the study over the next 3 - 6 months, such as severe medical or psychiatric disease, such as treatments for cancer or congestive heart failure, OR a condition that may require hospitalization or surgery
* Self-reported history of drowsy driving or fallen asleep while driving
* Night shift worker
* Prior exposure to Cognitive Behavioral Therapy for Insomnia (CBT-I) treatment
* Insomnia severity index score < 12

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | 6-8 weeks
  Mean change in Insomnia Severity Index (ISI) score from baseline to end of intervention. Score ranges from 0 to 28, with higher scores indicating a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No